CLINICAL TRIAL: NCT02186613
Title: Telephone Support From Primary Care to Breastfeeding Mothers: A Randomized and Multicenter Clinical Trial
Brief Title: Telephone Support From Primary Care for Breastfeeding Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4R14/015
Record Dates: First submitted 2014-06-29; First posted 2014-07-10 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Breast Feeding
Keywords: Breast Feeding; Telephone; Education; Primary Health Care
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): These mothers and their babies will receive Primary Care standard care (office visits at 1, 2, 4 and 6 months) plus the telephone support
  Interventions: Behavioral: Telephone support
- No intervention (No Intervention): Standard care (office visits at 1, 2, 4 and 6 months)

INTERVENTIONS:
Behavioral: Telephone support — Telephone support intervention to improve breastfeeding rates. The intervention will consist in weekly calls during the first two months and every two weeks between the second and the sixth month. The intervention will be done by pediatric nurses and we have developed a protocol of important issues to deal depending on the age of the baby.
  Arms: Experimental

SUMMARY:
The investigators will conduct a telephone-based support to breastfeeding women with healthy newborns to improve breastfeeding outcomes.

DETAILED DESCRIPTION:
The World Health Organization recommends exclusive breastfeeding to infants until 6 months of age in order to achieve optimum growth. The proportion of exclusive breastfeeding mothers at 6 months is only 24.7 in Spain. The investigators believe it is important to increase the proportion of breastfeeding mothers in their population. Therefore, the investigators have developed a telephonic support protocol for mothers. The intervention will be performed by pediatric nurses in Primary Care.

The main aim of this study is to evaluate in a randomized controlled trial the effectiveness of telephone-based breastfeeding support in exclusive breastfeeding. The secondary aim is to evaluate the effectiveness of the telephonic support in any breastfeeding.

The investigators hypothesis is that this intervention will increase exclusive breastfeeding and any breastfeeding rates.

The study will be carried out in Cornellà, a semi-urban area near Barcelona. Participants will include breastfeeding women who have full-term healthy infants. Mothers will be recruited upon their first arrival to Primary Care from hospital. Eligible mothers who consent to participate will be randomized into either the intervention group or the control group. The latter will receive standard postpartum care. The former will receive standard postpartum care, plus a weekly telephone call during the first two months and every 2 weeks thereafter between the second and the sixth month. The pediatric nurse responsible for monitoring the standard care of each and every patient will be the one responsible for contacting them via telephone. Therefore, the study is not blinded.

The evolution of exclusive breastfeeding will be compared to artificial or supplemented feeding at 1, 2, 4 and 6 months. The effect of the intervention on breastfeeding supplemented with formula will also be valued. Classification into breastfeeding categories is based on 24-hour dietary recall.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with healthy newborns
* 37 weeks gestation or greater
* Exclusive breastfeeding or any breastfeeding when arrive at Primary Care

Exclusion Criteria:

* Infant or mother admitted in ICU
* Twin pregnancy
* Major congenital malformation of babies
* Mothers age <= 18
* Inability to understand Spanish/Catalan
* Mothers who don't have a telephone
* Mothers who don't give her consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Rate of exclusive breastfeeding | 6 months
  Exclusive breastfeeding at 6 months. (time frame: 6 months)

SECONDARY OUTCOMES:
Rate of exclusive breastfeeding | 4 months
  Exclusive Breastfeeding at 4 months. (time frame: 4 months)
Rate of exclusive breastfeeding | 2 months
  Exclusive breastfeeding at 2 months. (time frame: 2 months)
Rate of exclusive breastfeeding | 1 month
  Exclusive breastfeeding at 1 month. (time frame: 1 month)

OTHER OUTCOMES:
Rate of non exclusive breastfeeding | 6 months
  Breastfeeding (non exclusive) at 6 months. (time frame: 6 months)
Rate of non exclusive breastfeeding | 4 months
  Breastfeeding (non exclusive) at 4 months. (time frame: 4 months)
Rate of non exclusive breastfeeding | 2 months
  Breastfeeding (non exclusive) at 2 months. (time frame: 2 months)
Rate of non exclusive breastfeeding | 1 month
  Breastfeeding (non exclusive) at 1 month. (time frame: 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Balaguer, Doctor, Principal Investigator — Jordi Gol i Gorina Foundation
Locations (1):
- Jordi Gol i Gurina Foundation, Barcelona, Barcelona, Spain